CLINICAL TRIAL: NCT03035968
Title: Improvement of Postural Control and Motor Function by Vojta Therapy in Early Stroke Rehabilitation of Stroke Patients - a Pilot Study and New Approach in Stroke Rehabilitation
Brief Title: Vojta Therapy in Early Stroke Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corina Epple (Other)
Responsible Party: Sponsor-Investigator, Corina Epple, Principle Investigator, Klinikum Frankfurt Höchst
Organization: Klinikum Frankfurt Höchst (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Höchster Vojta Stroke Studie
Record Dates: First submitted 2017-01-24; First posted 2017-01-30 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Vojta Therapy; Reflex Locomotion
Keywords: Vojta therapy; reflex locomotion; stroke rehabilitation; stroke; physiotherapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessor for the secondary outcome (Barthel Index and mRS after 90 days) is blinded. All other outcome assessors have knowledge of the interventions assigned to individual participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vojta arm (Experimental): Patients in the interventional arm are treated with Vojta therapy from randomization until discharge.
  Interventions: Other: Vojta therapy
- conventional physiotherapy arm (Active Comparator): Patients in this control arm are treated with conventional physiotherapy for motor improvement from randomization until discharge.
  Interventions: Other: conventional physiotherapy

INTERVENTIONS:
Other: Vojta therapy
  Other Names: reflex locomotion
  Arms: Vojta arm
Other: conventional physiotherapy
  Arms: conventional physiotherapy arm

SUMMARY:
Stroke is the major cause for permanent disability in adults. It is still unclear, which physiotherapeutic approaches are most effective. The Bobath-concept is one of the most widely used approaches in stroke rehabilitation within the western world, although several studies have failed to demonstrate superiority and showed partially even inferiority compared to other physiotherapy approaches. The Vojta therapy is based on a completely different approach - the reflex locomotion. However to date no study has been performed for stroke. We designed a randomized clinical trial (RCT) to compare Vojta and conventional physiotherapy in patients with acute ischemic (AIS) or hemorrhagic stroke (ICH). This RCT will be the first trial to investigate improvement of postural control due to Vojta therapy in early rehabilitation of stroke patients, which is a very new approach in stroke-rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (> 18 years)
* CT or MRI proven acute ischemic (AIS) or hemorrhagic stroke (ICH) within 72h after onset of symptoms
* Severe hemiparesis (medical research council scale for muscle strength ≤2)
* premorbid modified Rankin Scale (mRS) ≤3
* maximal National Institute of Health Stroke Scale Score (NIHSS) 25
* Voluntary written consent by the patient

Exclusion Criteria:

* Severe cognitive impairment due to aphasia or dementia, prohibiting that physiotherapeutic challenges can be understood.
* Participation on another clinical trial
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-12-02 (Actual); Primary Completion 2017-04-14 (Actual); Study Completion 2017-07-04 (Actual)

PRIMARY OUTCOMES:
Improvement of postural control measured with the trunc control test (TCT) on day 9 after admission to the hospital | Day 1-9 after admission to hospital (+/- 1)
  The Trunc Control Test (TCT) is a valid test to asses motor impairment after stroke. A range of 0 to 100 points can be achieved. Patients are tested before the first treatment on day 2, after 5 days and after the last intervention on day 9 (+/-1) after admission to hospital.

SECONDARY OUTCOMES:
Improvement of neglect measured with the Catherine Bergego Scale (part 5 and 6) after on day 9 after admission to the hospital (compared to baseline) | Day 1-9 after hospital admission (+/- 1)
  The neglect is assessed with part 5 and 6 of the Catherine Bergego Scale. Patients are tested before and after the first treatment on day 2, before and after treatment after 5 days and before and after the last intervention on day 9 (+/-1) after admission to hospital.
Improvement of arm motor function measured with the motor evaluation scale for upper extremity in stroke patients [MESUPES, part 1 to 4] on day 9 after admission to the hospital (compared to baseline) | Day 1-9 after hospital admission (+/- 1)
  The arm motor function is assessed with part 1 to 4 of the MESUPES. Patients are tested before and after the first treatment on day 2, before and after treatment after 5 days and before and after the last intervention on day 9 (+/-1) after admission to hospital.
Improvement of the Barthel Index on day 9 after admission to the hospital | Day 1-9 after hospital admission (+/- 1)
  The Barthel Index is assessed before the first treatment on day 2 and after the last intervention on day 9 (+/-1) after admission to hospital.
Improvement of the NIHSS on day 9 after admission to the hospital | Day 1-9 after hospital admission (+/- 1)
  The NIHSS is assessed before the first treatment on day 2 and after the last intervention on day 9 (+/-1) after admission to hospital.
Improvement of the neglect (measured with the Catherine Bergego Scale) before and after every single intervention. | Day 1-9.
  Patients are assessed for the neglect 3 times: on day 2, day 5 and day 9 (plus/minus 1 day) after admission to hospital before and after treatment. We want to compare if there is an improvement of the neglect directly after treatment.
Improvement of arm motor function (measured with the MESUPES) before and after every single intervention. | Day 1-9.
  Patients are assessed for the motor function 3 times: on day 2, day 5 and day 9 (plus/minus 1 day) after admission to hospital before and after treatment. We want to compare if there is an improvement of motor function directly after treatment.
Improvement of the modified Rankin Scale (mRS) on day 90 after stroke onset | Day 90 after stroke onset
  The mRS is assessed before the first treatment on day 2 after admission to hospital (before treatment) and on day 90 after stroke onset. The 90 day mRS is assessed via telephone interview by a blinded assessor
Improvement of the Barthel Index on day 90 after stroke onset | Day 90 after stroke onset
  The Barthel Index is assessed before the first treatment on day 2 after admission to hospital (before treatment) and on day 90 after stroke onset. The 90 day Barthel Index is assessed via telephone interview by a blinded assessor

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum Frankfurt Höchst, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Epple C, Maurer-Burkhard B, Lichti MC, Steiner T. Vojta therapy improves postural control in very early stroke rehabilitation: a randomised controlled pilot trial. Neurol Res Pract. 2020 Aug 20;2:23. doi: 10.1186/s42466-020-00070-4. eCollection 2020. PMID 33324926
- See also: Homepage of the International Vojta Society — http://www.vojta.com